CLINICAL TRIAL: NCT04486521
Title: Clinical Outcome of Anti-IL6 and Corticosteroid Monotherapy vs Combination in COVID-19 Cytokine Release Syndrome
Brief Title: Anti-IL6 and Corticosteroid Monotherapy vs Combination in COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Collaborators: Society of Critical Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: RAC # 2201053
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Critical Illness; Corona Virus Infection; Cytokine Release Syndrome
MeSH Terms: conditions — Critical Illness; Coronavirus Infections; Cytokine Release Syndrome | interventions — Interleukin-6; tocilizumab; siltuximab; Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental: anti-IL-6 drugs (tocilizumab and siltuximab)
  Interventions: Drug: Interleukin 6 (IL6) Antagonist
- Active Comparator 1: Anti-IL-6 drugs (tocilizumab and siltuximab) and corticosteroids combination
  Interventions: Drug: Interleukin 6 (IL6) Antagonist and corticosteroids
- Active Comparator 2: corticosteroids alone
  Interventions: Drug: corticosteroid alone

INTERVENTIONS:
Drug: Interleukin 6 (IL6) Antagonist — anti-IL6 alone
  Other Names: Tocilizumab; Siltuximab
  Groups: Experimental
Drug: Interleukin 6 (IL6) Antagonist and corticosteroids — anti-IL6 + corticosteroid combination
  Groups: Active Comparator 1
Drug: corticosteroid alone — dexamethasone, hydrocortisone, methylprednisolone, prednisone. All steroids " other than dexamethasone" will be converted to dexamethasone equivalent
  Groups: Active Comparator 2

SUMMARY:
The cytokine storms mediated by over production of proinflammatory cytokines have been observed in a large population of critically ill patients infected with COVID-19. Patients diagnosed with cytokine storms progress to cardiovascular collapse, multiple organ dysfunction and death rapidly. Therefore, early identification, treatment and prevention of the cytokine storms are of crucial importance for the patients. Immuomedulator such as interleukin-6 (IL-6) antagonist, emerged as an alternative treatment for COVID-19 patients with a risk of cytokine storms recently. In this study, we aimed to evaluate the safety and efficacy of anti-IL6 alone vs anti-IL6 corticosteroid combination in patients with COVID-19 pneumonia

DETAILED DESCRIPTION:
This study will provide further insight whether anti-IL6 alone provide same efficacy and clinical outcome with reasonable side effects profile compared to anti-IL6 + corticosteroid and might serve as a corticosteroid sparing agents in COVID-19 patient with cytokine storms. Data elements will be retrieved from VIRUS registry which is a prospective, non-interventional, multi-center, multi-national observational cross sectional study

ELIGIBILITY:
Inclusion Criteria:

1. Adult Critically ill patients
2. COVID-19 PCR positive
3. Presence of clinical and radiological signs of progressive disease, and laboratory evidence indicative of risk for cytokine storm complications.
4. Received anti-IL6 or corticosteroids as part of COVID-19 treatment

Exclusion Criteria:

1. Non COVID-19 related admissions
2. Repeated Admission to ICUs/Hospital
3. Patient did not receive anti-IL6 or corticosteroids

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data elements will be retrieved from Viral Infection and Respiratory Illness Universal Study: COVID-19 (VIRUS registry ClinicalTrials.gov Identifier: NCT04323787) which is a prospective, non-interventional, multi-center, multi-national observational cross sectional study.
Sampling Method: Probability Sample
Enrollment: 860 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-07-22 (Estimated); Study Completion 2021-07-22 (Estimated)

PRIMARY OUTCOMES:
Ventilator-Free Days | Up to Day 28
  The median ventilator-free days will be calculated as calendar days with no ventilator support to day 28 . Participants who die before day 28 are assigned zero free days.

SECONDARY OUTCOMES:
Median duration of ventilation | Up to Day 28
  From Intubation to extubation date and off Mechanical Ventilation or until ICU discharge, death, or 28 days whichever occurs first.
Median change in the PaO2/FiO2 | Up to Day 28
  Ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2)
Vasopressor-Free days | Up to Day 28
  The median vasopressor-free days will be calculated as calendar days with no vasopressor support to day 28. Participants who die before day 28 are assigned zero free days.
Duration of ICU Stay | Up to 28 days
  To compare ICU LOS
Duration of Hospital Stay | Up to 28 days
  To compare hospital LOS
Mortality Rate | Up to Day 28
  Death that occurs during 28 days
Percentage of participants with adverse events [transaminitis, hyperglycemia] | Up to 28 days
  adverse events that occurs during 28 days
Concentration of Ferritin, IL6, D dimer, fibrinogen, C-reactive protein (CRP), Lactate dehydrogenase (LDH) and absolute lymphocyte count and their correlation with the effectiveness of the treatment | Up to 28 days
  Concentration of inflammatory markers
Rate of superinfection (bacterial, viral, invasive fungal infections) | Up to 28 days
Time to the first COVID 19 test negative | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Amer, PharmD,BCPS, BCCCP, Principal Investigator — King Faisal Specialist Hospital and Research Center- Riyadh; Mohammed Bawazeer, MD,FRCSC,FACS, Principal Investigator — King Faisal Specialist Hospital and Research Center- Riyadh
Locations (1):
- King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Walkey AJ, Kumar VK, Harhay MO, Bolesta S, Bansal V, Gajic O, Kashyap R. The Viral Infection and Respiratory Illness Universal Study (VIRUS): An International Registry of Coronavirus 2019-Related Critical Illness. Crit Care Explor. 2020 Apr 29;2(4):e0113. doi: 10.1097/CCE.0000000000000113. eCollection 2020 Apr. PMID 32426754
- [Derived] Amer M, Kamel AM, Bawazeer M, Maghrabi K, Butt A, Dahhan T, Kseibi E, Khurshid SM, Abujazar M, Alghunaim R, Rabee M, Abualkhair M, Al-Janoubi A, AlFirm AT, Gajic O, Walkey AJ, Mosier JM, Zabolotskikh IB, Gavidia OY, Teruel SY, Bernstein MA, Boman K, Kumar VK, Bansal V, Kashyap R; Society of Critical Care Medicine Discovery Viral Infection and Respiratory Illness Universal Study (VIRUS): COVID-19 Registry Investigator Group. Clinical characteristics and outcomes of critically ill mechanically ventilated COVID-19 patients receiving interleukin-6 receptor antagonists and corticosteroid therapy: a preliminary report from a multinational registry. Eur J Med Res. 2021 Oct 2;26(1):117. doi: 10.1186/s40001-021-00591-x. PMID 34600589